CLINICAL TRIAL: NCT04601077
Title: Pilot Study: The Evaluation of Nitric Oxide Generating Lozenges on Outcome in Newly Diagnosed COVID-19 Patient of African American and Hispanic Origin
Brief Title: The Evaluation of Nitric Oxide Generating Lozenges on Outcome in Newly Diagnosed COVID-19 Patient of African American and Hispanic Origin
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study stopped due to futility.
Sponsor: Nitric Oxide Innovations LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IND150758 Pilot
Record Dates: First submitted 2020-10-21; First posted 2020-10-23 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Placebo Control
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide (Active Comparator): Nitric Oxide (NO) lozenges taken twice daily by mouth for 30 days
  Interventions: Drug: Nitric Oxide lozenges, 30 mg
- Placebo (Placebo Comparator): Placebo of Nitric Oxide (NO) lozenges taken twice daily by mouth for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide lozenges, 30 mg — Nitric Oxide lozenge, 30 mg twice a day for 30 days
  Arms: Nitric Oxide
Drug: Placebo — Placebo for Nitric Oxide lozenge, 30 mg twice a day for 30 days
  Arms: Placebo

SUMMARY:
This study is a multi-center, randomized, double blinded, prospective, placebo controlled study. Patients upon diagnosis of COVID-19 (Corona Virus Disease-19) will be eligible to participate in the study. The purpose of this study is to find out the side effects and ability to take the study drug, Nitric Oxide (NO) lozenges when taken twice daily by mouth. If this study shows that the drug has no or few, acceptable side effects, it will then include up to 840 participants to find out if the drug can reduce bad outcomes of COVID-19 infection (hospitalization, ICU admission, death). In each part of the study, half of the subjects will receive the study drug and the other half will be given a placebo (inactive pill).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of 50-85 years of age
2. Subjects with recent COVID-19 diagnosis (within 72 hours), that are symptomatic (fever, cough, SOB, weakness, or other flu-like symptoms).
3. Agrees to comply with study procedures (diary, oximeter readings, telephone follow up).
4. Has given voluntary, written, informed consent to participate in the study.
5. Identifies as African American or Hispanic Origin
6. Patients must have at least 1 risk factor (history of hypertension (BP> 140/99) CHF, angina, prior MI, coronary angiography with one significantly occluded vessel, diabetes mellitus, obesity, or smoking, (for at least 5 years).

Exclusion Criteria:

1. Females who are pregnant, breastfeeding or planning to become pregnant during the course of the study.
2. Patients unresponsive or unable to take anything by mouth (NPO).
3. Individuals who are cognitively impaired and/or who are unable to give informed consent.
4. Blood pressure below 110 mmHg systolic and 60 mmHg diastolic on entry into study.
5. History of syncope or other symptoms of orthostatic hypotension.
6. History of methemoglobinemia.
7. Severe case of G6PD deficiency

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation
Enrollment: 524 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Low blood pressure | 30 days
  Blood pressure under 90 mmHg
dizziness | 30 days
  Incidence of self reported dizziness

SECONDARY OUTCOMES:
Incidence of hospitalization, ICU admission, intubation, dialysis and death | 30 Days
  The effects of NO therapy on incidence of hospitalization, intubation, ICU admission, dialysis and death in treated patients vs. those receiving placebo therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- American Institute of Therapeutics, Lake Bluff, Illinois, United States

IPD SHARING:
Plan to Share IPD: No